CLINICAL TRIAL: NCT04427540
Title: Oxytocin Pharmacokinetics After Intramuscular Injection
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not initiated; no subjects were consented or enrolled
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00065842
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis, Knee
Keywords: advanced knee arthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Single IM injection of Oxytocin 17 micrograms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Oxytocin (Experimental): Single IM injection Oxytocin 17 micrograms
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin 10 micrograms IM
  Other Names: Pitocin

SUMMARY:
In this study people with knee arthritis so severe that a joint replacement is needed are recruited for a one day study. Study participants will have an intravenous catheter (IV) inserted in the forearm. A single intramuscular (IM) injection of oxytocin (Pitocin®), 17 micrograms will be administered and blood samples will be taken several times over the next 120 minutes. The amount of oxytocin will be measured in the blood samples.

The main purpose of this study is to sample the blood, before and after the administration of oxytocin and calculate the pharmacokinetics (amount of oxytocin in the blood over time) of oxytocin.

DETAILED DESCRIPTION:
This is an unblinded, sequential study of subjects, all will receive an intramuscular (IM) injection oxytocin with blood samples taken thereafter in order to create a formula to describe the concentrations of oxytocin in the blood over time (pharmacokinetics). In this study people with knee arthritis so severe that a joint replacement is needed are recruited for a one day study. Participants will come to the Clinical Research Unit (CRU) and have an intravenous catheter (IV) inserted in the forearm. Participants will get a single IM injection of oxytocin (Pitocin®), 17 micrograms (10 International Units (IU)) and blood will be taken several times over the next 120 minutes and the amount of oxytocin measured in the blood samples. This information will be analyzed by another group at Stanford University in the pharmacokinetics/pharmacodynamics (PK/PD) Core part of this application. The Core group at Stanford will use mathematics to fit the amount of oxytocin over time as it disappears from blood to a formula, called pharmacokinetics. The effect of subject age, sex, race, ethnicity and weight on the pharmacokinetics of oxytocin will be tested for, since these things can affect how quickly drugs circulate in the blood and are important to better adjust the dose of drug to the individual.

The main purpose of this study is to sample the blood and calculate the pharmacokinetics of oxytocin. The research participants will not benefit from this study, but the knowledge investigators get will be important not only to adjust oxytocin dose to individuals, but to study its possible effects on pain in a very standardized way. The sample size chosen is needed to get an accurate estimate for the parameters in the pharmacokinetic model for the population, not just the subjects in this study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female > 18 and < 75 years of age, Body Mass Index (BMI) <40.
* 2. Generally in good health as determined by the Principal Investigator based on prior medical history, American Society of Anesthesiologists physical status 1, 2, or 3.
* 3. Normal blood pressure or, for those with hypertension, pressure controlled with anti-hypertensives and with a resting heart rate 45-100 beats per minute.
* 4. Female subjects of child-bearing potential and those < 1 year post-menopausal, must be practicing highly effective methods of birth control such as hormonal methods (e.g., combined oral, implantable, injectable, or transdermal contraceptives), double barrier methods (e.g., condoms, sponge, diaphragm, or vaginal ring plus spermicidal jellies or cream), or total abstinence from heterosexual intercourse for a minimum of 1 full cycle before study drug administration.
* 5. diagnosis of advanced knee arthritis

Exclusion Criteria:

* 1. Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
* 2. Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (active gynecologic disease in which increased tone would be detrimental e.g., uterine fibroids with ongoing bleeding), compromise the subject's compliance with study procedures, or compromise the quality of the data
* 3. Women who are pregnant (positive result for serum pregnancy test at screening visit), women who are currently nursing or lactating, women that have been pregnant within 2 years
* 4. Subjects with neuropathy, chronic pain, diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Oxytocin concentration in serum | 1 minute post administration to 120 minutes post administration
  Amount of Oxytocin in serum measured in picograms/millilitres (pg/ml) after IM Oxytocin administered

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No